CLINICAL TRIAL: NCT07309367
Title: Web-based Advance Care Planning Intervention for Patients With Kidney Failure on Dialysis: Pilot Testing of 'My Voice'
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Duke-NUS Graduate Medical School (Other)
Collaborators: National Kidney Foundation, Singapore (Other)
Responsible Party: Principal Investigator, Chandrika Ramakrishnan, Research Fellow, Duke-NUS Graduate Medical School
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: NUS-IRB-2024-713
Record Dates: First submitted 2025-09-23; First posted 2025-12-30 (Actual); Last update posted 2025-12-30 (Actual); Status verified 2025-11

CONDITIONS: Kidney Failure, Chronic Therapy; Hemodialysis
Keywords: Advance care planning; Web intervention; Dialysis withdrawal
MeSH Terms: conditions — Renal Insufficiency

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group (Experimental): Patients will view My Voice website intervention and complete patient module. They will also receive standard of care for advance care planning [namely serious illness conversation (SIC)] with the health care provider at the dialysis centers.
  Caregivers will view My Voice website intervention and complete caregiver module.
  Interventions: Other: My Voice website intervention with patient and caregiver modules
- Usual care group (No Intervention): Patients will receive standard of care for advance care planning -namely the serious illness conversation (SIC) with the health care provider at the dialysis centres.
  Caregivers will receive no intervention.

INTERVENTIONS:
Other: My Voice website intervention with patient and caregiver modules — 'My Voice' is an interactive web-based ACP intervention tailored for patients with kidney failure on dialysis, and their caregivers, and includes patient and caregiver modules. Patient module has 6 steps consisting of a series of videos, value-clarification exercise (VCE) identifying goals and values for care, and knowledge quiz, and a summary My Voice document that is generated shared with patients, designated surrogates and HCPs. Automated reminders are sent to revisit My Voice. Caregiver module has 4 steps with videos and quiz, with access to their loved one's summary My Voice document containing goals of care and values.
  Arms: Intervention group

SUMMARY:
'My Voice' is a website intervention developed to enable advance care planning (ACP) conversations for patients with kidney disease on dialysis, educate patients on their illness, help identify their goals and preferences for EOL care, and coaches them on how to speak with their HCPs and loved ones. This study aims to evaluate if 'My Voice' intervention improves quality of ACP conversations between patients and providers, and patients and family carers; improves patient's knowledge about kidney failure, engagement in ACP and preparedness for future end of life care compared to usual practices for ACP in dialysis centres.

ELIGIBILITY:
Inclusion Criteria: For patients

* Singapore citizens or permanent residents; aged 21 years (age of majority) or older
* CKD stage 5; receiving dialysis
* Identified as eligible for SIC by NKF HCPs based on one or more of the following:

  1. clinical deterioration with a terminal condition or
  2. intolerability to dialysis or
  3. having two or more unplanned hospitalizations for renal complications in the past 6 months (from medical records); or
  4. known to palliative care or under conservative care as indicated in the discharge summary or
  5. poor functional status indicated by the Fragility Assessment for Elders (FIFE) score >4
* Normal cognitive function as indicated by Mini Mental Scale Examination (MMSE) score of 24 or more (based on medical record)
* Able to speak and read English, Mandarin or Malay
* Agreeable to be audio-recorded

Inclusion Criteria: For caregivers

* Aged 21 years old and above
* Family caregivers of the patients recruited i.e. Caregiver primarily involved in providing care, ensuring provision of care, and/or in making decisions regarding patient's care, with no expectation of financial compensation
* Able to speak and read English, Mandarin or Malay
* Have a phone and/or an electronic device with internet access.
* Agreeable to be audio-recorded

Exclusion Criteria: For Patients

* Patients with cognitive impairment or serious mental illness will be excluded
* Patients who had prior serious illness conversations (SIC) will be excluded
* Are not easily contactable via mobile phone or landline

Exclusion Criteria: For Caregivers

* Those who are foreign domestic workers/maids
* Are not easily contactable via mobile phone or landline

Min Age: 21 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2025-10-02 (Actual); Primary Completion 2026-09-30 (Estimated); Study Completion 2026-12-30 (Estimated)

PRIMARY OUTCOMES:
Quality of ACP conversations (serious illness conversations) between patients and physicians/health care providers | Post baseline and within 8 weeks
  Quality of ACP conversations will be measured using a scoring sheet developed for the study. One point will be given for every SICG topic discussed with score min to max of 0 to 13. Higher scores indicate higher quality.

OTHER OUTCOMES:
Change in kidney disease and dialysis knowledge scores | Baseline to 8 weeks
  Collected using knowledge questions designed by the research team. Higher scores indicate higher knowledge
Change in ACP engagement | Baseline to 8 weeks
  Using the 9-item Advance care planning engagement scale. 9 to 45 (Min to Max) value, with higher value indicating higher engagement
Change in patient preparedness | Baseline to 8 weeks
  Assessed using Preparedness for end-of-life decision-making scale. 20 to 80 (min to max) scores, with higher scores indicating better preparedness
Change in proportion of patients who had ACP conversations with family caregivers/spokesperson | Baseline and 8 weeks
  Based on self-reported number of ACP conversations collected in the survey

CONTACTS AND LOCATIONS:
Locations (1):
- Duke NUS Medical School, Singapore, Singapore

IPD SHARING:
Plan to Share IPD: No